CLINICAL TRIAL: NCT04441190
Title: A Novel, Digital, and Interactive Multi-mode Stroke Rehabilitation System of Arm and Hand: Development and Validation of Clinical Efficacy
Brief Title: Multi-mode Stroke Rehabilitation System: Development and Validation of Clinical Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201901885A3
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Cerebrovascular Disorders; Central Nervous System Diseases
Keywords: stroke; multi-mode rehabilitation; action observation; mirror therapy; digital image technology
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Action Observation Therapy (Digital AOT) (Experimental): The common categories of motor actions and tasks will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movement or object manipulation, and (c) upper-limb functional tasks.
  Interventions: Behavioral: Digital Action Observation Therapy (Digital AOT)
- Digital Mirror Therapy (Digital MT) (Experimental): The common categories of motor actions and tasks will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movement or object manipulation, and (c) upper-limb functional tasks.
  Interventions: Behavioral: Digital Mirror Therapy (Digital MT)
- Conventional Occupational Therapy (Active Comparator): The common categories of motor actions and tasks will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movement or object manipulation, and (c) upper-limb functional tasks.
  Interventions: Behavioral: Conventional Occupational Therapy

INTERVENTIONS:
Behavioral: Digital Action Observation Therapy (Digital AOT) — The participants will be asked to observe videos and then practice what the participants observed.
  Arms: Digital Action Observation Therapy (Digital AOT)
Behavioral: Digital Mirror Therapy (Digital MT) — The participants will observe the real-time self-recorded visual illusion, and move their upper limbs as could as possible.
  Arms: Digital Mirror Therapy (Digital MT)
Behavioral: Conventional Occupational Therapy — The participants will receive upper-limb training without providing videos for observing neither providing them mirror illusions of movements.
  Arms: Conventional Occupational Therapy

SUMMARY:
The specific study aims will be:

1. To develop the novel, digital, and interactive MSR system of arm and hand with integrated digital action observation therapy (AOT) and mirror therapy (MT).
2. To pilot usability testing for examining the feasibility of this new MSR system from the users' experiences and feedback.
3. To examine the treatment effects of digital AOT, digital MT and a control intervention in patients with stroke by conducting a randomized controlled trial.
4. To identify who will be the possible good responders to digital AOT and MT based on their baseline motor function and mental imagery abilities.

DETAILED DESCRIPTION:
Phase I: Multi-mode stroke rehabilitation (MSR) System Development & Usability Testing

Ten patients with stroke and 4 certified occupational therapists were recruited in this phase I study. During the pilot testing, each stroke patient will try to use each training mode of digital AOT and MT by the assistance of the therapist. At the end of the pilot testing, the patients and the therapists will be asked to complete the System Usability Scale and a self-designed questionnaire to assess the user experience and perspective about this new MSR system and their view of its suitability for stroke patients.

Phase II: Validation of Clinical Treatment Efficacy

This three-arm, single-blind, randomized controlled trial will investigate the treatment effects among the 3 groups of digital AOT, digital MT, and dose-matched control intervention. An estimated 60 patients with stroke will be recruited to participate in this phase II study. Each participant will receive a total of 15 training sessions (60 minutes per session) for 3 to 4 weeks. Clinical outcome measures will be conducted at baseline, immediately after treatment (the fourth week), and at 1 month follow-up after treatment.

ELIGIBILITY:
Phase I: Multi-mode stroke rehabilitation (MSR) System Development and Usability Testing

For stroke patients

Inclusion Criteria:

* diagnosed as having a unilateral stroke;
* aged from 20 to 80 years;
* a baseline score of the Fugl-Meyer Assessment in a range of 20 to 60;
* able to follow the instructions and able to provide user feedback verbally;
* without aphasia and neglect

For therapists

Inclusion Criteria:

* holding an occupational therapist license

Phase II: Validation of Clinical Treatment Efficacy

Inclusion Criteria:

* diagnosed as having a unilateral stroke;
* at least 6 months after stroke onset;
* aged from 20 to 80 years;
* a baseline score of FMA in a range of 20 to 60;
* able to follow the study instructions;
* capable of participating in therapy and assessment sessions

Exclusion Criteria:

* global or receptive aphasia,
* severe neglect,
* major medical problems or comorbidities that have influenced upper-limb usage or caused severe pain

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Meyer Assessment | baseline, 4 weeks, 2 months
  The upper-limb subsection of Fugl-Meyer Assessment is a measure with sound psychometric properties to evaluate motor impairments.
Change scores of Movement Imagery Questionnaire-Revised, Second Edition | baseline, 4 weeks, 2 months
  The Movement Imagery Questionnaire-Revised, Second Edition is a 14-item questionnaire with sound reliability and validity to evaluate the ability of motion imagination in patients with stroke.

SECONDARY OUTCOMES:
Change scores of Chedoke Arm and Hand Activity Inventory | baseline, 4 weeks, 2 months
  The Chedoke Arm and Hand Activity Inventory is a reliable and validated measure to assess the independence of stroke patients to perform activities of daily living with an affected upper limb.
Change scores of Box and Block Test | baseline, 4 weeks, 2 months
  The Box and Block Test is a tool with sound reliability and validity to evaluate hand dexterity of stroke patients.
Change scores of Revised Nottingham Sensory Assessment | baseline, 4 weeks, 2 months
  The Revised Nottingham Sensory Assessment is a standardized measure with good reliability to assess sensory function in patients with stroke.
Change scores of Barthel Index | baseline, 4 weeks, 2 months
  The Barthel Index is a validated tool designed to measure activities reflecting the daily living independence.
Change scores of Motor Activity Log | baseline, 4 weeks, 2 months
  The Motor Activity Log is a semi-structured interview with good psychometric properties to assess the level of use of affected upper limb in 30 main activities of daily living.
Change scores of the health state of EQ-5D-5L | baseline, 4 weeks, 2 months
  The questionnaire of EQ-5D-5L contains 5 dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and uses a 5-point Likert scale scored from 1 (no problem) to 5 (unable to/extreme problems); whereas, the numerical description of 5 dimensions represents the health state.
Change scores of the visual analogue scale (VAS) of EQ-5D-5L | baseline, 4 weeks, 2 months
  The VAS of EQ-5D-5L scores will be scored from 0 to 100, with a higher score indicating better overall current health.
Change of joint angles of OPAL wearable sensors | baseline, 4 weeks, 2 months
  The OPAL wearable sensors is used to objectively record the movements of an affected upper limb in patients with stroke in real time, such as joint angles. Joint angles of the shoulder, elbow, and wrist will be calculated.
Change of joint velocity of OPAL wearable sensors | baseline, 4 weeks, 2 months
  The OPAL wearable sensors is used to objectively record the movements of an affected upper limb in patients with stroke in real time, such as joint velocity. The angular velocity of shoulder, elbow, and wrist will be also collected.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wei Hsieh, PhD, Principal Investigator — Department of Occupational Therapy, College of Medicine, Chang Gung University
Locations (2):
- Taiwan (2):
  - Taipei Hospital, Ministry of Health and Welfare, New Taipei City
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh YW, Lee MT, Hsu YC, Wu KY, Chen CC. Digital Mirror Therapy and Action Observation Therapy for Chronic Stroke: A Pilot Randomized Controlled Trial. Occup Ther Int. 2025 Mar 20;2025:8741362. doi: 10.1155/oti/8741362. eCollection 2025. PMID 40151488